CLINICAL TRIAL: NCT06600659
Title: A Pilot Study to Establish Incidence and Characteristics of Patients at Risk for Symptomatic Hyperammonemia Secondary to Recombinant Erwinia Asparaginase
Brief Title: A Study to Determine Number of Patients Who Develop High Ammonia Levels After Receiving Recombinant Erwinia Asparaginase
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-006011; NCI-2024-01023 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-006011 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Acute Lymphobkastic Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood sample collection, complete surveys, and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates the incidence of symptomatic hyperammonemia (high ammonia levels) in patients being treated with recombinant Erwinia asparaginase.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine incidence of patients who develop hyperammonemia secondary to recombinant Erwinia asparaginase.

II. To characterize patients at risk for hyperammonemia secondary to recombinant Erwinia asparaginase.

OUTLINE: This is an observational study.

Patients undergo blood sample collection, complete surveys, and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Followed by pediatric hematology/oncology
* Receiving recombinant Erwinia asparaginase for treatment of malignancy

Exclusion Criteria:

* Patients < 1 year of age
* Patients who have previously received recombinant Erwinia asparaginase within the past two weeks

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving recombinant Erwinia asparaginase for treatment of malignancy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of patients who develop hyperammonemia | Up to 12 months
  Assessed by measuring ammonia levels via blood test. Baseline ammonia level will be determined around the time of consent. During the first two recombinant Erwinia asparaginase (Rylaze®) courses, there will be two blood draws per week. Each course of recombinant Erwinia asparaginase (Rylaze®) lasts for two weeks, so there will be four blood draws per course.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E. Martin, PharmD, RPh, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials